CLINICAL TRIAL: NCT07330050
Title: Phase II Clinical Trial Evaluating Whole Agonist-Stimulated T (WAST) Cells in Combination With Docetaxel as a Second-line Treatment for Advanced Non-small Cell Lung Cancer (NSCLC) Resistant to PD-1 Inhibitors
Brief Title: WAST Cell-Docetaxel Combination Therapy in PD-1 Inhibitor-Resistant Advanced NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20251324
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cell Count; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WAST Cells Plus Docetaxel (Experimental): Patients will receive WAST cells in combination with docetaxel once every 3 weeks for 4 cycles. Following completion of the combination phase, patients will continue on docetaxel monotherapy until disease progression, unacceptable toxicity, or voluntary withdrawal from the study.
  Interventions: Biological: Whole Agonist-Stimulated T (WAST) cells injection; Drug: Docetaxel

INTERVENTIONS:
Biological: Whole Agonist-Stimulated T (WAST) cells injection — WAST cells (≥4.0 × 10⁹ cells), intravenous infusion, d14, Q3W for 4 cycles.
Drug: Docetaxel — 75 mg/m², intravenous infusion, day 1, Q3W.

SUMMARY:
This prospective Phase II study aims to evaluate the preliminary efficacy and safety of WAST cells combined with docetaxel as second-line therapy in patients with advanced NSCLC resistant to PD-1 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* At screening, patients must meet the following diagnostic and treatment criteria: 1) Histologically or cytologically confirmed NSCLC, 2) Advanced NSCLC as determined by imaging according to AJCC V8, 3) Disease progression after first-line treatment with a PD-1 inhibitor; Expected survival time greater than 3 months;
* At screening, measurable target lesions on imaging with the longest diameter greater than 1.0 cm;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 at screening;
* Adequate bone marrow reserve at screening, defined as:

Absolute neutrophil count (ANC) >1.5×10⁹/L; Absolute lymphocyte count (ALC) ≥0.3×10⁹/L; Platelets (PLT) ≥100×10⁹/L; Hemoglobin (HGB) ≥100g/L;

* Adequate organ function at screening, meeting the following criteria:

Aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal (ULN) (≤5 ULN if due to tumor infiltration); Alanine aminotransferase (ALT) ≤2.5 times ULN (≤5 ULN if due to tumor infiltration); Total serum bilirubin ≤1.5 times ULN (≤3 ULN if due to tumor infiltration); Serum creatinine (Scr) ≤1.5 times ULN, or creatinine clearance rate ≥60 mL/min; Minimum lung reserve level, defined as ≤Grade 1 dyspnea and oxygen saturation >91% without supplemental oxygen; International Normalized Ratio (INR) ≤1.5 times ULN, and activated partial thromboplastin time (APTT) ≤1.5 times ULN;

* Women of childbearing potential must have a negative urine pregnancy test, and any male or female patient capable of having children must agree to use effective contraception throughout the study and for at least 1 year after the last dose of study treatment.

Exclusion Criteria:

* Patients with symptomatic central nervous system (CNS) metastases at screening (patients with asymptomatic CNS metastases, or those who have been treated locally and are stable without symptoms for 4 weeks, are eligible);
* History of CNS disorders prior to screening, such as epilepsy, cerebrovascular ischemia/hemorrhage, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar diseases, organic brain syndromes, psychiatric disorders, or any autoimmune diseases affecting the CNS;
* Received immunotherapy, targeted therapy, chemotherapy, or radiotherapy within 4 weeks before screening, and deemed unsuitable for enrollment by the investigator;
* Discontinued systemic corticosteroid therapy less than 72 hours before cell infusion; however, physiological replacement doses of steroids (e.g., prednisone <10 mg/day or equivalent) are allowed;
* Any history of adoptive cell therapy prior to screening;
* History of organ/tissue transplantation prior to screening;
* Known active systemic autoimmune diseases under treatment prior to screening;
* At screening, meets any of the following criteria:

Hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) positive; Hepatitis B e antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab) positive, with HBV-DNA copy numbers above the lower limit of quantification; Hepatitis C antibody (HCV-Ab) positive; Treponema pallidum antibody (TP-Ab) positive; HIV antibody test positive; EBV-DNA, CMV-DNA copy numbers above the lower limit of quantification;

* Undergone major surgery within 4 weeks prior to screening and deemed unsuitable for enrollment by the investigator;
* History of other malignancies within the past 2 years (except successfully treated non-melanoma skin cancer or in situ carcinoma);
* At screening, meets any of the following cardiac conditions:

Left ventricular ejection fraction (LVEF) ≤50% (by ECHO); New York Heart Association (NYHA) class III or IV congestive heart failure; Uncontrolled hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) or pulmonary hypertension despite standard treatment; Myocardial infarction or cardiac surgery within 12 months prior to cell infusion; Clinically significant valvular heart disease;

* Tumor involvement of the atrium or ventricle at screening;
* History of pulmonary interstitial fibrosis or severe chronic obstructive pulmonary disease (COPD);
* Presence of clinical emergencies requiring urgent intervention due to tumor obstruction or compression (e.g., bowel obstruction or vascular compression) at screening;
* Active bleeding at screening;
* History of deep vein thrombosis or pulmonary embolism within 6 months prior to screening;
* Vaccinated with live vaccines within 6 weeks prior to screening;
* Active infection requiring treatment at screening;
* Participation in another interventional clinical study within 4 weeks prior to screening;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Time Frame: Up to 24 months
  ORR was defined as the percentage of patients with a confirmed complete (CR) or partial response (PR) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  PFS was defined as the time from the initial treatment to the first occurrence of disease progression or all-cause death (whichever occurs first) assessed by the investigator according to RECIST v1.1.
Overall Survival (OS) | up to 3 years
  OS was defined as the time from the initial treatment until the date of death due to any cause.
Disease Control Rate (DCR) | up to 24 months
  DCR was defined as the proportion of patients with the best overall response of CR, PR, and stable disease (SD) as determined by the investigator according to RECIST 1.1.
Duration of response (DOR) | up to 24 months
  DOR was defined as first documented evidence of a CR or PR until PD or death as determined by the investigator according to RECIST v1.1.
Number of Participants Who Experienced an Adverse Event (AE) | up to 24 months (Serious AEs: Up to 90 days after last dose of study treatment (Other AEs: Up to 30 days after last dose of study treatment)
  An AE was defined as any untoward medical occurrence in a study participant administered with study drug and which does not necessarily have to have a causal relationship with this study drug. The number of participants who experienced an AE is presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No